CLINICAL TRIAL: NCT07256899
Title: Comparison of Transversus Fascial Plane Block and Anterior Quadratus Lumborum Block for Lower Urogenital Surgery in Pediatric Patients.
Brief Title: Analgesic Comparison of Transversus Fascial Plane and Quadratus Lumborum Blocks in Pediatric Urogenital Procedures
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Münevver Kayhan, Lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ctf-qlb/tfpb-02
Record Dates: First submitted 2025-11-20; First posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Regional Anesthesia Block; Anesthesia and Analgesia; Pediatric Anesthesia; Pediatric Regional Anesthesia
Keywords: anterior QLB; Transversalis Fasia Plane block; Pediatric Regional Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dental Occlusion

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment design in which participants are randomly allocated to one of two intervention groups: the Anterior Quadratus Lumborum Block (QLB) group or the Transversalis Fascia Plane (TFP) block group. Each participant receives only one type of block, and there is no crossover between groups. Randomization is performed using a computer-generated sequence with allocation concealment. Postoperative pain evaluators and data analysts are blinded to the group assignments.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded to the type of block they receive. The anesthesiologist performing the block is aware of the assignment due to the nature of the intervention. Postoperative pain assessments and data analysis will be conducted by personnel blinded to the treatment groups to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior QLB - Preoperative ultrasound-guided anterior quadratus lumborum block (Experimental): Preoperative ultrasound-guided anterior quadratus lumborum block administered according to standardized anesthesia protocol.
  Interventions: Procedure: Anterior Quadratus Lumborum Block (QLB)
- TFP Block - Preoperative ultrasound-guided transversalis fascia plane block (Experimental): Preoperative ultrasound-guided transversalis fascia plane block administered according to standardized anesthesia protocol.
  Interventions: Procedure: Transversalis Fascia Plane (TFP / TAP) Block

INTERVENTIONS:
Procedure: Anterior Quadratus Lumborum Block (QLB) — Participants in this group will receive a preoperative ultrasound-guided anterior quadratus lumborum block. The block will be performed under sterile conditions using an in-plane technique with a linear ultrasound probe. The dose of 0.4 ml/kg of 0.25% bupivacaine will be administered according to age and weight. Standardized anesthesia protocols will be applied for all patients. Postoperative pain will be assessed using FLACC scores, and additional analgesics will be administered if required.
  Arms: Anterior QLB - Preoperative ultrasound-guided anterior quadratus lumborum block
Procedure: Transversalis Fascia Plane (TFP / TAP) Block — Participants in this group will receive a preoperative ultrasound-guided transversalis fascia plane block. The block will be performed supine under sterile conditions using an in-plane technique with a linear ultrasound probe. The dose of 0.4 ml/kg of 0.25% bupivacaine will be administered according to age and weight. Standardized anesthesia protocols will be applied for all patients. Postoperative pain will be assessed using FLACC scores, and additional analgesics will be administered if required.
  Arms: TFP Block - Preoperative ultrasound-guided transversalis fascia plane block

SUMMARY:
This study aims to compare the analgesic effectiveness of the preoperatively administered Anterior Quadratus Lumborum Block (Anterior QLB) and the Transversalis Fascia Plane Block (TFP block) in children undergoing lower abdominal urogenital surgery. The study will include children aged 6 months to 12 years, with randomization performed using the sealed opaque envelope method, and outcome assessment conducted in a double-blinded manner. All patients will receive a standardized anesthesia protocol, and the regional blocks will be performed under ultrasound (US)-guided techniques.

Perioperative evaluations will include pain levels, hemodynamic responses, additional analgesic requirements, block performance time, technical success rate, and family satisfaction. Postoperative pain will be monitored using the Face, Legs, Activity, Cry, Consolability (FLACC) scale, and analgesics will be administered when necessary. By comparing these two commonly used regional anesthesia techniques, this study aims to contribute to improved perioperative pain management strategies in the pediatric population.

DETAILED DESCRIPTION:
Regional anesthesia techniques have become increasingly preferred in pediatric anesthesia due to their ability to enhance multimodal analgesia, reduce opioid use and associated side effects, and potentially prevent the development of chronic pain (1). With the widespread adoption of ultrasonography (USG), peripheral nerve blocks have gained popularity as safer alternatives to central neuraxial blocks, which carry a higher complication risk. Truncal blocks have become particularly important in abdominal surgeries. Various quadratus lumborum block (QLB) approaches have demonstrated the ability to provide extensive sensory blockade (T4-L2 dermatomes) in cadaveric and clinical studies. However, because the number of randomized controlled trials in this area remains limited, further research is needed to better establish the efficacy of QLB (2).

The anterior quadratus lumborum block (Anterior QLB) provides effective analgesia for procedures such as inguinal hernia repair and orchiopexy, likely due to its potential spread toward the paravertebral space. The transversalis fascia plane (TFP) block provides analgesia by anesthetizing the ilioinguinal and iliohypogastric nerves as they travel along the ventral surface of the quadratus lumborum muscle and course between the transversalis fascia and the transversus abdominis muscle. These nerves originate from the anterior ramus of the L1 spinal nerve, with contributions from T12.

The primary aim of this study is to compare the effects of the TFP block and the Anterior QLB, performed preoperatively, on perioperative pain levels and analgesic requirements in pediatric patients undergoing lower abdominal urogenital surgery. Secondary aims include evaluating postoperative pain, additional analgesic needs, hemodynamic responses, block performance times, technical success rates, and patient and family satisfaction.

Methods:

Children aged 6 months to 12 years scheduled for inguinal hernia repair or orchiopexy will be enrolled. Exclusion criteria include allergy to local anesthetics, infection at the injection site, coagulopathy or other contraindications to regional anesthesia, inability to obtain informed consent, planned laparoscopic orchiopexy, American Society of Anesthesiologists (ASA) physical status class IV, and anticipated postoperative intensive care requirements.

Randomization will be performed using a sealed opaque envelope method, and outcome assessment will be double-blinded. Following premedication, all participants will undergo standard monitoring, including electrocardiography (ECG), peripheral oxygen saturation (SpO₂), and non-invasive blood pressure (NIBP) measurement. Anesthesia induction will be performed with thiopental, fentanyl, and rocuronium, followed by intubation; maintenance anesthesia will be achieved with sevoflurane.

Participants will be allocated into two groups:

Group 1: Anterior Quadratus Lumborum Block (Anterior QLB)

Group 2: Transversalis Fascia Plane Block (TFP block)

All blocks will be performed under sterile conditions using a linear ultrasound transducer and an in-plane technique with appropriately sized (18-22 gauge) intravenous cannulas. All patients will receive 0.4 mL/kg of 0.25% bupivacaine.

Perioperative monitoring will include recording the block-to-incision duration and heart rate (HR) and blood pressure (BP) measurements at baseline and at 5, 10, 20, 30, 45, and 60 minutes after incision. If additional analgesia is required, remifentanil infusion will begin at 0.1 mcg/kg/min and be titrated in response to hemodynamic changes.

Postoperatively, patients will be monitored for 2 hours in the recovery unit and then transferred to the pediatric surgery ward. Pain will be assessed using the Face, Legs, Activity, Cry, Consolability (FLACC) scale, and patients with a FLACC score of ≥4 will receive acetaminophen and/or tramadol. Families will receive information regarding postoperative pain management, and structured telephone follow-up will be conducted at 16 and 24 hours to evaluate family satisfaction, which will be recorded on a 3-point scale (1 = not satisfied, 2 = partially satisfied, 3 = very satisfied).

This study aims to compare the analgesic efficacy of two regional anesthesia techniques widely used in pediatric urogenital surgery and to contribute to the development of safer and more effective perioperative pain management strategies in children.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 months to 12 years
* Scheduled for lower abdominal urogenital surgery (e.g., inguinal hernia repair, undescended testis surgery)
* ASA physical status I-III
* Parental/guardian informed consent obtained

Exclusion Criteria:

* Allergy to local anesthetics
* Infection at the injection site
* Coagulopathy or other contraindications to regional anesthesia
* Laparoscopic orchiopexy scheduled
* ASA physical status IV
* Inability to obtain consent from parent/guardian
* Expected need for postoperative intensive care

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain Score | 0, 5, 10, 20, 30, 45, 60 minutes intraoperatively; 2, 4, 8, 12, 24 hours postoperatively
  Pain intensity will be assessed using the FLACC scale (Face, Legs, Activity, Cry, Consolability) at predefined time points. The primary outcome is the difference in perioperative pain levels between the Anterior Quadratus Lumborum Block (QLB) and Transversalis Fascia Plane (TFP) block groups.

SECONDARY OUTCOMES:
Total Analgesic Consumption | First 24 hours postoperatively
  Total amount of analgesics (including remifentanil, tramadol, and paracetamol) administered within 24 hours will be recorded and compared between groups.
Time to First Rescue Analgesia | 0-24 hours postoperatively
  Time from the end of surgery to the first additional analgesic administration will be measured.
Parent/Patient Satisfaction | 16th and 24th postoperative hours
  Parents will be contacted by phone to assess satisfaction with pain management using a 3-point Likert scale (1 = not satisfied, 2 = partially satisfied, 3 = very satisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Kendigelen, Principal Investigator — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Munevver Kayhan, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty; Ayse Cigdem Tutuncu, Professor Doctor, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty
Locations (1):
- Istanbul University-Cerrahpasa, Cerrahpasa Medicine of Faculty, Bakırköy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No